CLINICAL TRIAL: NCT01081535
Title: The Effect of IV PCA With Ketorolac or Fentanyl Combined With Caudal Block for Postoperative Analgesia in Small Children Undergoing Intravesical Ureteroneocystostomy
Brief Title: The Effect of Intravenous (IV) Patient Controlled Analgesic (PCA) With Ketorolac or Fentanyl Combined With Caudal Block for Postoperative Analgesia in Small Children Undergoing Intravesical Ureteroneocystostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Kil Hae Keum/professor, Yonsei University, College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2009-0107
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-01

CONDITIONS: Ureteroneocystostomy
Keywords: Pediatric patients (6 months-5 years) scheduled elective ureteroneocystostomy
MeSH Terms: interventions — Ketorolac; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketorolac (Experimental)
  Interventions: Drug: ketorolac, fentanyl
- fentanyl (Experimental)
  Interventions: Drug: ketorolac, fentanyl

INTERVENTIONS:
Drug: ketorolac, fentanyl — intravenous PCA

SUMMARY:
The effect of IV PCA with ketorolac or fentanyl combined with caudal block for postoperative analgesia in small children undergoing intravesical ureteroneocystostomy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled for elective ureteroneocystostomy were enrolled.

Exclusion Criteria:

* History of allergy to aspirin or NSAIDs
* Peptic ulcer disease, and renal function impairment.
* And local infection foci on back, spinal anomalies
* Infectious diseases
* Neurologic disorders
* Seizures and coagulopathies were excluded for sacral epidural block.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Children's Hospital of Eastern Ontario Pain Scale, CHEOPS and Faces, Legs, Activity, Cry, and Consolability, FLACC | postoperative 24 hours, 48hours

CONTACTS AND LOCATIONS:
Overall Officials: Hae Keum Kil, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea